CLINICAL TRIAL: NCT06279078
Title: Long-term Comparative Effectiveness for Osteoporosis/Osteoporosis and Metabolic Disease in Adult Asthmatic Patients Maintaining Inhaled/Systemic Corticosteroid: a Real-world Evidence
Brief Title: Long-term Effect of Steroid on Metabolic Diseases in Asthmatics
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Hyun-Seob Jeon, Clinical fellow, dept. of Allergy and Clinical Immunology, Ajou University School of Medicine
Other Study IDs: AJOUIRB-DB-2023-446
Record Dates: First submitted 2024-01-10; First posted 2024-02-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Asthma; Osteoporosis, Osteopenia; Osteoporosis Risk; Osteoporotic Fractures
Keywords: asthma; osteoporosis; corticosteroid; inhaled corticosteroid; fractures
MeSH Terms: conditions — Asthma; Osteoporosis; Bone Diseases, Metabolic; Osteoporotic Fractures; Fractures, Bone | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Corticosteroid — oral/inhaled corticosteroid
  Other Names: inhaled corticosteroid

SUMMARY:
The goal of this retrospective/observational study is to compare the clinical outcomes between the high-cumulative-dose group and the low- cumulative-dose group of oral/inhaled corticosteroid in the long-term management of asthma patients. The main hypothesis are:

i. High cumulative dose of corticosteroid is related to the prevalence of osteoporosis/osteoporosis in the long-term management of adult asthma.

ii. High cumulative dose of corticosteroid can affect populations that have a high-risk of osteoporosis (females over 50 years of age).

iii. High cumulative dose of corticosteroid is related to the prevalence of diabetes mellitus, hypertension, and hyperlipidemia in the long-term management of adult asthma.

iv. High cumulative dose of corticosteroid affects bone metabolism-related diagnostic tests and laboratory values and the prescription rate of bone metabolism-related medications.

ELIGIBILITY:
A. Inclusion criteria i. Adult asthmatics (over 18 years) who have maintained inhaled corticosteroid with or without systemic corticosteroid for more than 12 months before the index date in our Medical Center.

ii. At least 1 asthma diagnosis within 1 year before the first corticosteroid exposure date by asthma specialists at Ajou University Medical Center (AUMC, Suwon, South Korea) with informed consent.

iii. A high cumulative dose is defined as the dose of corticosteroids above the mean cumulative dose of corticosteroids prescribed during 1 year.

iv. The equivalent dose will use for calculating the mean cumulative dose of each inhaled corticosteroid inhaler or systemic corticosteroid prescribed.

v. Prescriptions within 365 days from the first prescription will be assumed to be continuous, and the cohort end date will be defined as the end of the continuous drug exposure.

B. Exclusion criteria i. Patients younger than 18 years ii. Patients younger than 50 years and males in high-risk population cohorts iii. Patients with osteoporosis or osteoporosis-related major fracture outcomes (pathological fracture due to osteoporosis, closed fracture of the femur, pelvis, and vertebral column) before the index date iv. Patients with corticosteroid-related outcomes (diabetes mellitus, hypertension, hyperlipidemia) before the index date (for secondary endpoint).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthma patients that visited AUMC (Ajou University Medical Center) from 1994 to 2023
Sampling Method: Probability Sample
Enrollment: 19968 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of osteoporosis/osteopenia | 5 years
  Prevalence of osteoporosis/osteopenia according to cumulative dose of steroid will be compared with incidence, incidence rate, and hazard ratio

SECONDARY OUTCOMES:
Bone mineral density (BMD) score | 5 years
  Change of BMD score (T-score), especially for L1-L4 and femur neck. (Z-score will also be evaluated for premenopausal women and men under 50 years of age)
Total alkaline phosphatase | 5 years
  Change of bone metabolism-related tests
Corrected calcium | 5 years
  Change of bone metabolism-related tests
Serum phosphate | 5 years
  Change of bone metabolism-related tests
Serum albumin | 5 years
  Change of bone metabolism-related tests (known to be reduced in osteoporosis patients)
prevalence of steroid related comorbidities(Diabetes Mellitus, Hypertension, Hyperlipidemia, etc.) | 5 years
  Compare the prevalence of steroid related comorbidities(Diabetes Mellitus, Hypertension, Hyperlipidemia, etc.) according to cumulative dose of steroid with incidence, incidence rate, and hazard ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Medical Center, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided